CLINICAL TRIAL: NCT05648851
Title: A Combination Retrospective and Prospective Natural History Study of Patients With Sanfilippo Syndrome Type D (MPSIIID)
Brief Title: A Natural History Study of Sanfilippo Syndrome Type D
Acronym: MPSIIID
Status: Completed | Type: Observational
Sponsor: Phoenix Nest (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: ALL-127; 1UB1NS122644-01A1 (NIH)
Record Dates: First submitted 2022-02-01; First posted 2022-12-13 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Sanfilippo Syndrome Type D
Keywords: Sanfilippo syndrome type D; mucopolysaccharidosis; MPSIIID
MeSH Terms: conditions — Mucopolysaccharidosis III; Mucopolysaccharidoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood (plasma and serum), cerebrospinal fluid (CSF), urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1 In person combination retrospective and prospective Natural History Study: Combination retrospective and prospective Natural History Study of patients living with Sanfilippo syndrome type D. The study will include home video of daily living activities via the RARE app, a mobile app designed for this study. In clinic visits will include neurocognitive, developmental, behavioral, biochemical, imaging measures as well as retrospective medical record analysis.
- Group 2 Retrospective medical record analysis: Retrospective collection and analysis of medical records of deceased or living patients.

SUMMARY:
Sanfilippo syndrome type D is a ultra rare syndrome with limited available natural history data. This study is planned to document, through retrospective and prospective data collection, syndrome progression in children and young adults with Sanfilippo syndrome type D. The results from this study may inform future clinical studies in targeted therapies for patients with Sanfilippo syndrome type D and may serve as an external control since there are very few patients with Sanfilippo syndrome type D.

DETAILED DESCRIPTION:
This is a single-center, natural history study of subjects with Sanfilippo syndrome type D. This study will combine a retrospective review of medical records and an ongoing collection of clinical data on an observational basis from participants with Sanfilippo syndrome type D.

Participants will be asked to attend clinic visits in person on a yearly basis. In clinic visits will include neurocognitive, developmental, behavioral, biochemical, imaging measures as well as retrospective medical record analysis. At 6-month intervals between clinic visits, participants will be contacted remotely for some safety assessments (e.g., collecting information about concomitant medications, concurrent illnesses, and procedure-related adverse events [AEs] and serious AEs [SAEs] since last clinic visit). At 6-month intervals, caregivers will complete questionnaires and record home video assessments using a dedicated, compliant study application (app) called RARE (Recording Application for Real-World Evidence). The RARE app consists of 9 tasks of Activities of Daily Living and socialization as well as two parent reported questionnaires.

No formal power or sample size calculations will be performed. At least 4 and up to 10 patients living with Sanfilippo syndrome type D will be enrolled in the prospective and retrospective study (group/cohort 1). An additional 5 patients deceased or living will be enrolled for retrospective medical record collection only (group/cohort 2).

The objectives of this study are:

1. To enhance the understanding of the natural history and progression of Sanfilippo syndrome type D.
2. To define and categorize clinical endpoints that may be used in future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in the study, patients must meet all of the following criteria:

1. Confirmed diagnosis of Sanfilippo syndrome type D disease by all of the following:

   1. Deficiency in alpha-GNS enzyme activity
   2. Has presented with signs/symptoms consistent with Sanfilippo syndrome type D, or, for individuals who have not presented with signs/symptoms of disease (eg, siblings of known patients), the determination of eligibility will be at the discretion of the Sponsor in conjunction with the site Investigator
   3. Genomic DNA analysis demonstrating homozygous or compound heterozygous, pathogenic and/or potentially pathogenic variants in the GNS gene
   4. Accumulated GAG HS in urine
2. Written informed consent from parent or legal guardian and assent from patient, if required
3. Parent/legal guardian willing to accompany the patient to all study visits
4. Ability to comply with protocol requirements, in the opinion of the Investigator
5. Negative urine pregnancy test at screening (nonsterile females of childbearing potential only) -

Exclusion Criteria:

Patients who meet any of the following criteria will not be eligible to participate in the study:

1. Have received an investigational drug within 30 days prior to the Baseline Visit
2. Concomitant illness or medical condition or extenuating circumstance that, in the opinion of the Investigator, might compromise the patient's ability to comply with protocol requirements, the patient's well-being or safety, or the interpretability of the patient's clinical data
3. The presence of significant non-MPS IIID-related CNS impairment or behavioral disturbances that would confound the scientific rigor or interpretation of results of the study -

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a documented diagnosis of Sanfilippo syndrome type D and who are currently untreated with investigational products (drugs/device) for this disease
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-01-22 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Cognitive function | Baseline, 12 months and 24 months
  Assessed using the Leiter-3, evaluation of nonverbal cognitive, neuropsychological abilities. The Leiter-3 emphasizes fluid intelligence a measure of the individuals innate cognitive abilities. Children's Color Trail Test (CCTT) assesses sustained attention, sequencing, and other executive functions while reducing reliance on language.
Change From Baseline in Motor function | up to 24 months
  Assessed using the MFM-32, 25 foot walk test in the clinic at baseline, 12 months and 24 months and video tasks via the RARE app task assessments: 'walking up/down stairs', 'transferring to sit' at baseline, 6 months, 12 months, 18 months and 24 months. Fine and gross motor skills will be assess at baseline, 6 months, 12 months, 18 months and 24 months via the RARE app task assessments: 'writing on paper', 'eating snack', 'looking at book', 'playing Uno', 'washing hands' and 'putting on jacket'.
Change From Baseline in Speech and language abilities | up to 24 months
  Assessed using the Preschool Language Scales Fifth Edition (PLS-5); parent reported questionnaire to be administered in the clinic at baseline, 12 months, 24 months. The PLS-5 is a comprehensive developmental language tool with questions that range from pre-verbal, interaction-based skills to emerging language to early literacy. Picture description is an informal speech tool used to analyze structural language skills, patients speech will be captured via the RARE app in the clinic at baseline, 12 months and 24 months. Expressive and receptive language abilities are embedded in several of the RARE app tasks: 'looking at book', 'playing Uno', 'putting on jacket' and will be captured at baseline, 6 months, 12 months, 18 months and 24 months.

SECONDARY OUTCOMES:
Change From Baseline in Functional abilities | up to 24 months
  Participants functional abilities will be captured via the RARE app at baseline, 6 months, 12 months, 18 months, 24 months while performing tasks of Activities of Daily Living (ADLs). ADLs include: Clothing Management, Eating and Drinking, Chewing and Swallowing, Hygiene, Maintaining and Changing positions, Writing Skills, and Walking. The Vineland Adaptive Behavioral Scales second addition (VABS-II) ia a parent reported clinical outcome assessment which will be administered in the clinic at baseline, 12 months and 24 months. The VABS-II Domains: Communication, Daily Living Skills, Socialization and Motor Skills will be used to assess patient's functional abilities.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Chung, MD, Principal Investigator — Columbia University Department of Pediatrics; Andres Morales, MD, Principal Investigator — Columbia University Department of Pediatrics
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
The data collected as part of the observational study may be analyzed and published. Phoenix Nest recognizes the importance of communicating medical study data and therefore encourages the publication of these data in reputable scientific journals and at seminars or conferences. The details of the processes of producing and reviewing reports, manuscripts, and presentations based on the data from this study will be described in the Clinical Trial Agreement between Phoenix Nest and the Investigator/institution. Consideration for authorship of all publications will be based on compliance with the Uniform Requirements for Manuscripts Submitted to Biomedical Journals ("Uniform Requirements") of the International Committee of Medical Journal Editors (http://www.icmje.org/ethical_1author.html) and Good Publication Practices.